CLINICAL TRIAL: NCT03799705
Title: Identifying Genetic Variants in Nicotinamide Adenine Dinucleotide (NAD) Synthesis Pathway in Patients With Congenital Malformations
Brief Title: Genetic Variants in Nicotinamide Adenine Dinucleotide (NAD) Synthesis Pathway
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Myra J. Wick, Principal Investigator, Mayo Clinic
Other Study IDs: 18-001135
Record Dates: First submitted 2018-08-29; First posted 2019-01-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Vacterl Association; Congenital Malformation
MeSH Terms: conditions — VACTERL association; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA and metabolites will be extracted from blood and urine for genetic variant and targeted metabolomics analyses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- History of VACTERL or congenital malformations: 1) Adults with VACTERL association; 2) adults with a history of congenital malformations resembling VACTERL association; 3) gravid and non-gravid women with a history of recurrent miscarriage, their surviving offspring, and the biological father of offspring; 4) newly diagnosed VACTERL patients identified by healthcare providers.

SUMMARY:
Researchers are trying to identify versions of genes as well as factors in subjects blood associated with certain types of congenital malformations(CMs). This study will help the researchers to better understand family traits that contribute to CMs.

ELIGIBILITY:
Inclusion Criteria:

1. Adults with confirmed or putative diagnosis of VACTERL association;
2. Families (mother, father, biological offspring) with a history of VACTERL-associated malformations
3. Gravid or non-gravid women with a history of miscarriage and/or offspring with non-VACTERL-associated malformations
4. Willingness to abstain from red meat, meat products, chicken, peanuts, or brewer's yeast (including beer) at least 24 hours prior to blood and urine collection

Exclusion Criteria:

1) Parents of non-biological children 3) Children with congenital malformations associated with an identifiable environmental or lifestyle exposure 4) Children with congenital malformations associated with confirmed chromosomal disorders 5) Failure to abstain from red meat, meat products, chicken, peanuts, or brewer's yeast (including beer) at least 24 hours prior to blood and urine collection.

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A US population consisting of adults with VACTERL, adults and offspring with a family history of VACTERL, and women with a history of miscarriage and/or congenital malformations.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Genetic variants | 2 years
  Identification of genetic variants which may be associated with VACTERL association or other congenital malformations.
Targeted metabolomics | 2 years
  Identification of changes in metabolic pathways which may provide functional insight into the presence of genetic variants in patients with VACTERL association

CONTACTS AND LOCATIONS:
Overall Officials: Myra Wick, MD PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials